CLINICAL TRIAL: NCT03619499
Title: Non Invasive Ventilation Versus Invasive Ventilation in Management of Bronchiolitis
Brief Title: Non Invasive Ventilation in Bronchiolitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Omran, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIVVIVIMOB
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Non Invasive Ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non invasive (Experimental): infants who fulfill criteria of severe bronchiolitis will be connected to non invasive ventilation
  Interventions: Device: non invasive ventilation
- invasive (No Intervention): infants who were connected to invasive mechanical ventilation

INTERVENTIONS:
Device: non invasive ventilation — patients who will fulfill the criteria of severe bronchiolitis will be connected to non invasive ventilation including continuous positive airway pressure via nasal prongs or nasal mask. Mode of ventilation, inspired oxygen levels, oxygen saturation, respiratory rate, and blood gas values from arterial samples prior to and after 2 and 4 hrs of ventilation or nearest time, will be documented.
  Arms: non invasive

SUMMARY:
It is decided to perform a prospective study in a non-selected population of infants with bronchiolitis during one year ( October.2018 to October.2019) to study the characteristics, clinical course and outcome of the use of Non invasive ventilation in the management and compare the results with those treated with invasive ventilation to assess safety and efficacy and inform guideline construction.

DETAILED DESCRIPTION:
Acute viral bronchiolitis is one of the most common respiratory diseases in early childhood and is a major health problem worldwide. The seasonal burden of the disease, the number of hospitalizations each year and the risk of subsequent asthma bring about substantial costs in developed countries. Respiratory syncytial virus and Human Rhinovirus seem to be the most frequent etiologic agents, but other viruses such as human Metapneumovirus, Influenza virus, and Parainfluenza virus can also be involved. The spectrum of clinical outcomes is wide, but bronchiolitis is more severe when caused by Respiratory syncytial virus. In contrast, while Human Rhinovirus is involved in milder forms, it is more likely to be associated with recurrent wheezing in infancy. Acute respiratory failure from pneumonia, influenza, and respiratory syncytial virus is responsible for 4.25 million deaths world-wide and the leading cause of mortality in low and middle-income countries. In the United Kingdom up to 7% of bronchiolitis admissions require intensive care for ventilatory support. One third of unplanned infant admissions to pediatric intensive care units have respiratory failure, the majority due to bronchiolitis, require invasive mechanical ventilation for 4-7 days and a prolonged hospital stay. In countries where there is no retrieval infrastructure, the need to develop safe and effective alternatives to invasive ventilation and pediatric intensive care unit admission is acute. However, none of the interventions commonly used for infants admitted with bronchiolitis is backed by robust evidence of benefit for clinically significant outcomes, making this a pressing subject for further study. Typically, intensive respiratory support for bronchiolitis is via invasive mechanical ventilation through an artificial airway, an intervention with recognized complications in infants. There is evidence to support the use of non-invasive ventilation in pediatric acute respiratory failure of variable causes.Although evidence for use in bronchiolitis is increasing,clinical acceptance is not universal and published best practice guidelines are not easily available.

ELIGIBILITY:
Inclusion Criteria:

* all infants with acute severe bronchiolitis,
* infants aged below 1 year.

Exclusion Criteria:

* patients who have contraindications for NIV (patients with maxillofacial trauma, gastrointestinal obstruction and severe secretion),
* Children who had suspected or confirmed underlying chronic diseases (i.e., cystic fibrosis, chronic pulmonary disease, congenital heart disease, bronchopulmonary disease, prematurity,
* Children who had already more than one wheezing episode.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
decrease risk of respiratory failure | 2 days
  in the form of ( pulse oximetry less than 94⁒, pao2 less than 60mmHg, paco2 more than 84mmHg ) while on NIV that lead to connection to invasive mechanical ventilation.

SECONDARY OUTCOMES:
decrease length of hospital stay | 7 days
  by prevention of ventilation acquired pneumonia and barotrauma that occur from use of invasive ventilation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andreola B, Bressan S, Callegaro S, Liverani A, Plebani M, Da Dalt L. Procalcitonin and C-reactive protein as diagnostic markers of severe bacterial infections in febrile infants and children in the emergency department. Pediatr Infect Dis J. 2007 Aug;26(8):672-7. doi: 10.1097/INF.0b013e31806215e3. PMID 17848876
- [Result] Feuillet F, Lina B, Rosa-Calatrava M, Boivin G. Ten years of human metapneumovirus research. J Clin Virol. 2012 Feb;53(2):97-105. doi: 10.1016/j.jcv.2011.10.002. Epub 2011 Nov 9. PMID 22074934
- [Result] Gern JE. The ABCs of rhinoviruses, wheezing, and asthma. J Virol. 2010 Aug;84(15):7418-26. doi: 10.1128/JVI.02290-09. Epub 2010 Apr 7. PMID 20375160
- [Result] Koponen P, Helminen M, Paassilta M, Luukkaala T, Korppi M. Preschool asthma after bronchiolitis in infancy. Eur Respir J. 2012 Jan;39(1):76-80. doi: 10.1183/09031936.00040211. Epub 2011 Jun 23. PMID 21700604
- [Result] Mathew JL. What works in bronchiolitis? Indian Pediatr. 2009 Feb;46(2):154-8. No abstract available. PMID 19242034
- [Result] Marguet C, Lubrano M, Gueudin M, Le Roux P, Deschildre A, Forget C, Couderc L, Siret D, Donnou MD, Bubenheim M, Vabret A, Freymuth F. In very young infants severity of acute bronchiolitis depends on carried viruses. PLoS One. 2009;4(2):e4596. doi: 10.1371/journal.pone.0004596. Epub 2009 Feb 25. PMID 19240806
- [Result] Midulla F, Pierangeli A, Cangiano G, Bonci E, Salvadei S, Scagnolari C, Moretti C, Antonelli G, Ferro V, Papoff P. Rhinovirus bronchiolitis and recurrent wheezing: 1-year follow-up. Eur Respir J. 2012 Feb;39(2):396-402. doi: 10.1183/09031936.00188210. Epub 2011 Aug 18. PMID 21852336
- [Result] Khilnani P, Singhi S, Lodha R, Santhanam I, Sachdev A, Chugh K, Jaishree M, Ranjit S, Ramachandran B, Ali U, Udani S, Uttam R, Deopujari S. Pediatric Sepsis Guidelines: Summary for resource-limited countries. Indian J Crit Care Med. 2010 Jan;14(1):41-52. doi: 10.4103/0972-5229.63029. PMID 20606908
- [Result] American Academy of Pediatrics Subcommittee on Diagnosis and Management of Bronchiolitis. Diagnosis and management of bronchiolitis. Pediatrics. 2006 Oct;118(4):1774-93. doi: 10.1542/peds.2006-2223. PMID 17015575
- [Result] Valkonen H, Waris M, Ruohola A, Ruuskanen O, Heikkinen T. Recurrent wheezing after respiratory syncytial virus or non-respiratory syncytial virus bronchiolitis in infancy: a 3-year follow-up. Allergy. 2009 Sep;64(9):1359-65. doi: 10.1111/j.1398-9995.2009.02022.x. Epub 2009 Mar 23. PMID 19416146
- [Result] Wainwright C, Altamirano L, Cheney M, Cheney J, Barber S, Price D, Moloney S, Kimberley A, Woolfield N, Cadzow S, Fiumara F, Wilson P, Mego S, VandeVelde D, Sanders S, O'Rourke P, Francis P. A multicenter, randomized, double-blind, controlled trial of nebulized epinephrine in infants with acute bronchiolitis. N Engl J Med. 2003 Jul 3;349(1):27-35. doi: 10.1056/NEJMoa022226. PMID 12840089
- [Result] Yanez LJ, Yunge M, Emilfork M, Lapadula M, Alcantara A, Fernandez C, Lozano J, Contreras M, Conto L, Arevalo C, Gayan A, Hernandez F, Pedraza M, Feddersen M, Bejares M, Morales M, Mallea F, Glasinovic M, Cavada G. A prospective, randomized, controlled trial of noninvasive ventilation in pediatric acute respiratory failure. Pediatr Crit Care Med. 2008 Sep;9(5):484-9. doi: 10.1097/PCC.0b013e318184989f. PMID 18679148
- [Result] Zorc JJ, Hall CB. Bronchiolitis: recent evidence on diagnosis and management. Pediatrics. 2010 Feb;125(2):342-9. doi: 10.1542/peds.2009-2092. Epub 2010 Jan 25. PMID 20100768